CLINICAL TRIAL: NCT02128451
Title: The Value of Adding Either Meperdine or Fentanyl to Clonidine-bupivacaine Mixture in Patients With Lower Limb Orthopedic Surgery Using Combined Spinal Epidural Anesthesia
Brief Title: The Value of Adding Either Meperdine or Fentanyl to Clonidine-bupivacaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman Abd Al-maksoud Yousef, assistant Professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 1350/14
Record Dates: First submitted 2014-04-06; First posted 2014-05-01 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Amputation Stumps
Keywords: meperdine ,fentanyl, clonidine, orthopedic surgery .
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Meperdine group (Active Comparator): 15ml 0.5% bupivacaine,25 mg of meperdine and 1 ml of clonidine will be injected epidurally in meperdine Group.
  Interventions: Drug: Meperdine
- Fentanyl group (Active Comparator): 15ml 0.5% bupivacaine, 25 micrograms of fentanyl and 1 ml of clonidine will be injected epidurally in fentanyl Group
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Meperdine — 15ml 0.5% bupivacaine,25 mg of meperdine and 1 ml of clonidine will be injected epidurally in meperdine Group.
  Other Names: Pethedine
  Arms: Meperdine group
Drug: Fentanyl — 15ml 0.5% bupivacaine, 25 micrograms of fentanyl and 1 ml of clonidine will be injected epidurally in fentanyl Group
  Other Names: fenta vera
  Arms: Fentanyl group

SUMMARY:
The use of clonidine as an alternative to epidural opioids offers several potential benefits. Clonidine does not have respiratory depressant effects, and the incidence of vomiting and pruritus is less frequent compared with that seen after administration of epidural morphine.

Epidural clonidine have focused on the optimal doses of clonidine to be used, rather than analyzing the potential advantage of using epidural clonidine versus opioids with respect to efficacy and incidence of side effects.

Epidural fentanyl has been used effectively as an alternative to morphine and has been shown to induce fewer complications when compared with epidural morphine. However, the incidence of vomiting in patients receiving epidural fentanyl still ranges between 28% and 52% depending on the study population and concentration used. The analgesic and side effects profile of epidural clonidine compared with epidural fentanyl are unknown.

The primary aim of this randomized double-blind trial is to test the hypothesis that epidural clonidine decreases the incidence of side effects compared with epidural fentanyl.

Therefore, we compared the hemodynamic effects of the epidural bupivacaine-clonidine- fentanyl combination with those of epidural bupivacaine- clonidine- meperdine. The secondary aim of this study was to determine the analgesic efficacy of bupivacaine-clonidine- fentanyl combination in comparison to bupivacaine- clonidine- meperdine combination.

DETAILED DESCRIPTION:
A prospective randomized double-blind clinical trial design was used in a cohort of ninety patients of both genders, physical status American Society of Anaesthesiologist (ASA) I and II who will undergo lower limb orthopedic surgery, will be enrolled into the present study.

Patients will divided randomly into two equal groups: Epidural Bupivacain-clonidine and fentanyl (BF) Group and Bupivacain-clonidine and meperdine (BM) Group, comprising of 45 patients each. Randomization will be performed by random numbers using sealed envelopes without sex stratification. Sealed envelopes indicate the group of assignment. An independent anesthesiologist, who did not participate in the study or data collection, will read the number contained in the envelope and made group assignments. Patients will be blindly randomized to the two groups; the process of inclusion into the study will go on until the requested number of patients will be reached.

Patients will be excluded from the study if their preoperative medication included opioid or non-opioid analgesics, corticosteroids, or non-steroidal anti-inflammatory drugs. Coagulation disorders, pregnancy, age less than 18 year, patient refusal, and emergency re-operation within the first 24hours also were exclusion criteria.

Under full aseptic conditions, the epidural space was identified at the L 2-3 or L 3-4 lumbar interspace using the loss-of-resistance to saline technique using 16-gauge Tuohy needle. An injection of 2 ml of hyperbaric bupivacaine will be injected into the subarachnoid space through 25 gauge spinal needle, then 15ml 0.5% bupivacaine, 25 micrograms of fentanyl and 1 ml of clonidine will be injected epidurally in fentanyl (F) Group, while 15ml 0.5% bupivacaine,25 mg of meperdine and 1 ml of clonidine will be injected epidurally in meperdine (M) Group.

The injection will be given with unlabelled syringes prepared by independent anaesthologist not involved in the patients care or in pain assessment. The specific treatment given is unknown to the patient, anesthesiologist, surgeon, or nurses in charge of pain assessment. All patients and personnel involved in patient management and data collection are unaware of the group to which the patient will be assigned.

On the evening before surgery, patients will be instructed about the use of a 10-cm visual analog scale (VAS) (0 = no pain to 10 = worst possible pain).

Postoperative pain will be assessed by independent physicians who will completely blinded to patients group assignment not sharing in the study design or data collection, visual analogue scale (VAS) ranging from 0 (no pain) to 10 (worst imaginable pain). Pain level will be recorded at PACU every 3 h for the first 24h. All patients received 15 mg/kg i.v. acetaminophen every 6 h; the first dose will be given 40 min before the end of surgery. Supplementary doses of acetaminophen i.v. will be given to patients with a VAS higher than 4. Any episodes of bradycardia (HR< 50 beats/min), hypotension (SBP< 90 mmHg), nausea, vomiting, and excessive sedation were recorded.

The primary outcome is the degree of postoperative pain score using VAS in the two groups. The secondary outcomes measures are analgesic requirement of the two groups during the first 24 h after surgery. All adverse events related to surgery and the regional anesthetic technique will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adults ASA I, II.
* Elective orthopedic lower limb surgery

Exclusion Criteria:

* Patients will be excluded from the study if their preoperative medication included opioid or non-opioid analgesics, corticosteroids, or non-steroidal anti-inflammatory drugs. Coagulation disorders, pregnancy, age less than 18 year, patient refusal, and emergency re-operation within the first 24hours also were exclusion criteria.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
the hemodynamic effects | 1 hour after epidural application
  the hemodynamic parameter (heart rate and blood pressure)

SECONDARY OUTCOMES:
the analgesic efficacy | 24 hours
  the analgesic efficacy using visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Ayman A Yousef, MD, Principal Investigator — Assistant Professor
Locations (2):
- Egypt (2):
  - Faculty of Medicine ,Tanta University., Tanta, Algharbiya
  - Tanta University Hospitals, Tanta, Algharbyia

REFERENCES:
- [Derived] Yousef AA, Atef AM, Awais WM. Comparison of fentanyl versus meperidine as supplements to epidural clonidine-bupivacaine in patients with lower limb orthopedic surgery under combined spinal epidural anesthesia. BMC Anesthesiol. 2015 Oct 14;15:146. doi: 10.1186/s12871-015-0126-5. PMID 26468074